CLINICAL TRIAL: NCT02274064
Title: Motivating Type O- Blood Donors to Return
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio University (Other)
Collaborators: New York Blood Center (Other); Hoxworth Blood Center (Other)
Responsible Party: Principal Investigator, Christopher R. France, Ph.D., Distinguished Professor, Ohio University
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: R56HL119180 (NIH)
Record Dates: First submitted 2014-10-21; First posted 2014-10-24 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Blood Donors
Keywords: Retention; Blood Donor Motivation
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Donors randomly assigned to this group will receive a motivational interview and implementation intention intervention telephone call.
  Interventions: Behavioral: Motivational Interview and Implementation Intention
- Control (No Intervention): Donors randomly assigned to this group will receive a standard donor recruitment telephone call.

INTERVENTIONS:
Behavioral: Motivational Interview and Implementation Intention — Telephone call that includes motivational interviewing techniques and develops an implementation intention plan.
  Arms: Intervention

SUMMARY:
This study develops a motivational interview and implementation intention intervention for blood donor retention and tests the efficacy of this new approach among first-time, Group O donors.

DETAILED DESCRIPTION:
In this study the investigators will recruit first-time Group O- and O+ donors four weeks after their donation using the donor databases of New York Blood Center and Hoxworth Blood Center. Eligible donors will be contacted via email and invited to participate in the study. Interested donors will be randomly assigned to either the Intervention condition where they will receive a motivational interview and implementation intention intervention phone call or to the Control condition where they will receive a standard donor recruitment phone call. Outcome measures will be assessed before and after the telephone contact using online questionnaires, and donation attempts will be tracked for one year. The investigators will use survival analysis to examine the effects of this intervention on retention during this one-year follow-up. Path analyses will also be used to examine potential mediators of the intervention effect. The investigators hypothesis is that donors who receive the motivational interview and implementation intention intervention will have larger increases in positive donation attitudes and perceived behavioral control which will contribute to enhanced intention and donation attempts.

ELIGIBILITY:
Inclusion Criteria:

* donor with New York Blood Center or Hoxworth Blood Center
* one previous donation
* O- or O+ blood
* eligible to donate again

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 598 (Actual)
Dates: Start 2014-11; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Repeat donation | 1 year from the date of next donor eligibility (i.e., 13 months post-intervention)
  number and timing of repeat donation attempts in one year following eligibility of donor return

SECONDARY OUTCOMES:
Donation attitude | 1 week pre- and 1 week post-intervention
  questionnaire
Donation subjective norm | 1 week pre- and 1 week post-intervention
  questionnaire
Donation perceived behavioral control | 1 week pre- and 1 week post-intervention
  questionnaire
Donation intention | 1 week pre- and 1 week post-intervention
  questionnaire
Donation decisional balance | 1 week pre- and 1 week post-intervention
  questionnaire
Donor identity | 1 week pre- and 1 week post-intervention
  questionnaire
Donation moral norm | 1 week pre- and 1 week post-intervention
  questionnaire
Donation anticipated regret | 1 week pre- and 1 week post-intervention
  questionnaire
Donation anxiety | 1 week pre- and 1 week post-intervention
  questionnaire
Donor self-efficacy (action and coping) | 1 week pre- and 1 week post-intervention
  questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Christopher R France, PhD, Principal Investigator — Ohio University
Locations (1):
- Ohio University, Athens, Ohio, United States